CLINICAL TRIAL: NCT03194698
Title: Pilot Study to Examine Efficacy and Cytokines Levels After Meibomian Gland Expression (MGX) With and Without Intense Pulsed Light Treatment (IPL)
Brief Title: Efficacy of IPL Treatment of Dry Eye and Ocular Rosacea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Joanne F. Shen, M.D., Chair, Department of Ophthalmology - Arizona, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16-008492
Record Dates: First submitted 2017-06-17; First posted 2017-06-21 (Actual); Results first posted 2020-01-03 (Actual); Last update posted 2020-01-03 (Actual); Status verified 2019-12

CONDITIONS: Ocular Rosacea; Dry Eye
Keywords: Intense Pulsed Light
MeSH Terms: conditions — Rosacea; Dry Eye Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- MGX and Intense Pulsed Light Treatment (IPL) (Experimental): Treatment with 4 visits and 4 treatments of IPL and Meibomian Gland Expression (MGX)
  Interventions: Device: Intense Pulsed Light Treatment (IPL); Procedure: Meibomian Gland Expression
- Meibomian Gland Expression (MGX) (Active Comparator): Treatment with 4 visits and 4 treatments of MGX only
  Interventions: Procedure: Meibomian Gland Expression

INTERVENTIONS:
Device: Intense Pulsed Light Treatment (IPL) — IPL is a high-intensity light source consisting of visible light in the wavelength range of 515-1200 nm, that is aimed at the eyes. Treatments are spaced four to six weeks apart for a total of 4 treatments.
  Arms: MGX and Intense Pulsed Light Treatment (IPL)
Procedure: Meibomian Gland Expression — Manual expression of the meibomian glands by placing the thumb against the lid margin and press firmly against the eyeball to determine the percentage of meibomian pores that are blocked. This assessment is performed on both the upper and lower lid of each eye.

SUMMARY:
Dry eye disease (DED) is a common condition that causes ocular discomfort and reduces visual acuity. The two categories of DED are evaporative dry eye and aqueous deficient dry eye. Both conditions can involve pathology of the meibomian glands, lacrimal glands, lids, tear film and surface cells. Meibomian gland dysfunction (MGD) is the leading cause of evaporative dry eye and contributes to aqueous deficient dry eye. The goal of MGD therapy is to provide long term improvement of symptoms for patients by improving the quality of meibum, increasing meibum flow, improving tear film stability and decreasing inflammation.

Commonly used therapies include preservative free drops, omega-3 fatty acid supplementation, topical cyclosporine, serum tears, topical azithromycin, oral doxycycline, moisture chambers, intraductal probing, lib margin exfoliation, automated thermal pulsation, warm compresses, among other. Despite this variety of symptoms, patients often do not experience complete or long term relief of symptoms.

Forced meibomian gland expression (MGX) has been shown to be an effective method of rehabilitating meibomian glands and improving dry eye symptoms. The eyelid margins are forcefully compressed to express gland contents. Research has shown improvement in patient symptoms with the use of MGX.

Intense pulsed light (IPL) have been used in dermatology to treat various conditions. Patients with DED who have tried other therapies and found no relief, often resort to IPL as a last resort. Research has shown IPL alone may be effective in improving patient symptoms. In addition, such studies have failed to show significant adverse events with the use of IPL.

Here, we propose a prospective, randomized, case controlled clinical pilot study to examine the efficacy for both subjective and objective measures. 20 patients with DED will be recruited and will be randomly assigned to one of two groups: MGX alone or MGX with IPL. Objective measures will include tear cytokine levels, impression cytology, meibography, tear osmolarity and others. Subjective measures will include quality of life screening tools.

We hypothesize that the use of MGX with IPL will lead to greater improvement in subjective dry eye symptoms and objective measures. Given the lack of adverse effects reported in the literature, we do not anticipate adverse effects in our study.

Rochester staff Drs. Faustch and Bourne are providing clinical research advice but have no contact with subjects or biospecimens.

ELIGIBILITY:
Dry eye of moderate severity with ocular rosacea diagnosed by ophthalmologist. No contraindications of severe ocular surface disease or inability to be safely treated with IPL.

Dry eye symptoms must be alleviated with topical anesthetic. No GVHD, Stevens Johnson, active allergic conjunctivitis or other conjunctivitis, alkali burn history.

Subjects must have at least 50% meibomian glands viable on meibography and no new treatments for dry eye in the past 6 months.

Contact lenses and refractive surgery is okay.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-08-17 (Actual); Primary Completion 2018-12-06 (Actual); Study Completion 2018-12-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joanne F Shen, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Arizona, Scottsdale, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sagaser S, Butterfield R, Kosiorek H, Kusne Y, Maldonado J, Fautsch MP, Patel D, Shen JF. Effects of Intense Pulsed Light on Tear Film TGF-beta and Microbiome in Ocular Rosacea with Dry Eye. Clin Ophthalmol. 2021 Jan 27;15:323-330. doi: 10.2147/OPTH.S280707. eCollection 2021. PMID 33536740
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | MGX and Intense Pulsed Light Treatment (IPL) | Meibomian Gland Expression (MGX)
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MGX and Intense Pulsed Light Treatment (IPL) | Meibomian Gland Expression (MGX) | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.3 (11.7) | 60.5 (12.1) | 59.9 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 10 | 17
  Male | 3 | 0 | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic/Latino | 0 | 1 | 1
  Not Disclosed | 1 | 0 | 1
  White | 9 | 9 | 18
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Change in Ocular Surface Disease Index (OSDI) Symptom Survey Score
Description: Symptom survey on severity of dry eye symptoms. This 12-item questionnaire assesses dry eye symptoms and the effects it has on vision-related function in the past week of the patient's life. The questionnaire has 3 subscales: ocular symptoms, vision-related function, and environmental triggers. Patients rate their responses on a 0 to 4 scale with 0 corresponding to "none of the time" and 4 corresponding to "all of the time." A final score is calculated which ranges from 0 to 100 with scores 0 to 12 representing normal, 13 to 22 representing mild dry eye disease, 23 to 32 representing moderate dry eye disease, and greater than 33 representing severe dry eye disease.
Time Frame: baseline, 3 months
Measure: Mean (Standard Deviation); unit: percentage of change in OSDI score
Arm/Group | MGX and Intense Pulsed Light Treatment (IPL) | Meibomian Gland Expression (MGX)
Number analyzed (Participants) | 10 | 10
percentage of change in OSDI score | -25.9 (20.0) | -2.0 (17.9)
Statistical Analysis 1: Comparison: MGX and Intense Pulsed Light Treatment (IPL) vs Meibomian Gland Expression (MGX); Test type: Superiority; p = 0.0312, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Change in Meibomian Glands Open - Right Lower Lid
Description: The count of manual expression of the meibomian glands. A thumb is placed against the lid margin and press firmly against the eyeball to determine the percentage of meibomian pores that are blocked. This assessment is performed on both the upper and lower lid of each eye.
Time Frame: baseline, 3 months
Measure: Mean (Standard Deviation); unit: percentage of blocked meibomian pores
Arm/Group | MGX and Intense Pulsed Light Treatment (IPL) | Meibomian Gland Expression (MGX)
Number analyzed (Participants) | 10 | 10
percentage of blocked meibomian pores | 6.9 (11.0) | 5.0 (11.0)
Statistical Analysis 1: Comparison: MGX and Intense Pulsed Light Treatment (IPL) vs Meibomian Gland Expression (MGX); Test type: Superiority; p = 0.79, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Change in Meibomian Glands Open - Left Lower Lid
Description: as for outcome 2
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: percentage of blocked meibomian
Arm/Group | MGX and Intense Pulsed Light Treatment (IPL) | Meibomian Gland Expression (MGX)
Number analyzed (Participants) | 10 | 10
percentage of blocked meibomian | 14.4 (16.1) | 10.0 (14.1)
Statistical Analysis 1: Comparison: MGX and Intense Pulsed Light Treatment (IPL) vs Meibomian Gland Expression (MGX); Test type: Superiority; p = 0.74, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: Adverse Events were collected over a period of 3 months
Arm/Group | MGX and Intense Pulsed Light Treatment (IPL) | Meibomian Gland Expression (MGX)
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-04-28): https://cdn.clinicaltrials.gov/large-docs/98/NCT03194698/Prot_SAP_000.pdf